CLINICAL TRIAL: NCT04103645
Title: A 2-tiered, Phase 2, Rule-based, Intra-patient Dose Escalation Study to Investigate Safety and Feasibility of Vactosertib (TEW-7197) in the Treatment of Anemic Patients With Philadelphia Chromosome-negative MPNs (Ph-neg MPNs)
Brief Title: Intra-patient Dose Escalation Study to Investigate Safety and Feasibility of Vactosertib in Treating Anemic MPN Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-06020285
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Anemia
MeSH Terms: conditions — Myeloproliferative Disorders; Anemia | interventions — vactosertib

STUDY DESIGN:
Intervention Model Description: This is an intra-patient dose finding study which starts with low dose of vactosertib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tier 1: Vactosertib 50 mg BID (Experimental): Vactosertib intra-patient dose finding cohort.
  Interventions: Drug: Vactosertib
- Tier 1: Vactosertib 100 mg BID (Experimental)
  Interventions: Drug: Vactosertib
- Tier 1: Vactosertib 150 mg BID (Experimental)
  Interventions: Drug: Vactosertib
- Tier 1: Vactosertib 200mg BID (Experimental)
  Interventions: Drug: Vactosertib
- Tier 2: Vactosertib (Experimental)
  Interventions: Drug: Vactosertib

INTERVENTIONS:
Drug: Vactosertib — 50 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
  Other Names: TEW-7197
  Arms: Tier 1: Vactosertib 50 mg BID
Drug: Vactosertib — 100 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
  Other Names: TEW-7197
  Arms: Tier 1: Vactosertib 100 mg BID
Drug: Vactosertib — 150 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
  Other Names: TEW-7197
  Arms: Tier 1: Vactosertib 150 mg BID
Drug: Vactosertib — 200 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
  Other Names: TEW-7197
  Arms: Tier 1: Vactosertib 200mg BID
Drug: Vactosertib — The lowest dose level of vactosertib for which no DLT was observed in Tier 1 AND The lowest dose level for which at least one of the 12 subjects enrolled on Tier 1 met Criteria for Clinical Benefit. Or, if a single dose level does not fulfil both Criterion 1 and Criterion 2, the starting dose level for Tier 2 will lowest dose from Tier 1 for which no DLT was identified.
  Other Names: TEW-7197
  Arms: Tier 2: Vactosertib

SUMMARY:
This study assesses the potential of using a TGFβ receptor inhibitor for the treatment of anemic patients with myeloproliferative neoplasms. TGFβ signaling is known to be abnormally high in patients with myeloproliferative neoplasms and it is thought that abnormal TGFβ signals cause many of the problems with blood cell formation in these diseases. The study design allows all patients to receive the study drug, vactosertib. The dose of vactosertib is individualized within a pre-set range based upon its effectiveness and tolerability. A total of up to 37 patients will be treated.

DETAILED DESCRIPTION:
This is a two-tiered multi arm Phase 2 trial of vactosertib (TEW-7197) for the treatment of anemia in Ph-neg MPNs. Both tiers use a rule-based, accelerated dose escalation scheme to efficiently assess the potential of vactosertib to safely and effectively treat anemic patients with Ph-neg MPNs. The first tier of this trial (Tier 1) is an intra-patient dose finding study in 12 patients that uses a low starting dose of vactosertib for all patients. Treatment dose is escalated according to prospectively-defined rules, and a toxicity and treatment effect algorithm during the period of 16 weeks (4 treatment cycles). If pre-established efficacy and safety endpoints are met, then Tier 1 of the study will be followed by a Tier 2 expansion study with an additional 25 patients for a period of 24 weeks (6 treatment cycles).

Vactosertib will be administered concurrently with the patient's current treatment (if any). Prior to enrollment, patients must be on a stable dose of their current therapy for 3 months prior to entering the study. Supportive care measures including packed red blood cell (PRBC) transfusions for HGB <7g/dL, or symptomatic anemia, will be permitted. Administration of erythropoiesis stimulating agents (ESAs), however, will not be permitted on the trial (patients recruited would have serum EPO >125 U/L above which the benefit of ESAs is not supported).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the WHO 2016 criteria for a Ph-neg MPN (including PV, ET, MF, MDS/MPN, MPN-U).

* Patients with MF must have DIPSS+ Intermediate or High-risk MF (primary of post-PV/ET).
* For patients receiving cytoreductive therapy, they should be on a stable dose of current cytoreductive therapy for at least 3 months prior to C1D1.
* Anemia as defined by HGB < 10 g/dL, or transfusion of ≥ 2 packed red blood cell (PRBC) unit within the past 4 weeks with HGB ≤8.5g/dL.
* Ineligible, unsuitable or refractoriness to ESA therapy defined as any of the following:

  * Serum erythropoietin (EPO) >125 U/L.
  * Proven ESA unsuitability is defined by history of any of the following:
  * Loss of erythroid hematologic improvement while receiving stable or increased ESA dose; or
  * ESA-attributed toxicity that, in the treating physician's opinion, makes ESA therapy unsuitable for subject.
  * ESA refractoriness defined by lack of erythroid hematologic improvement to ESA:27
  * Less than 1.5 g/dL increase in hemoglobin after at least 6 weeks of ESA therapy; or
  * Ongoing transfusion dependence that has not been reduced by > 4U over an 8-week period compared to ESA pre-treatment 8 weeks.
* Acceptable Cardiovascular status

Exclusion Criteria:

* Any other serious medical condition which in the Investigator's opinion would preclude safe participation in the study.
* Patients with history of TIA or stroke within the past 12 months are excluded.
* Female subjects who are breastfeeding, or intend to breastfeed, during the study or in the 30 days following the last dose of study drug are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Scandura, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez-Boluda JC, Correa JG, Garcia-Delgado R, Martinez-Lopez J, Alvarez-Larran A, Fox ML, Garcia-Gutierrez V, Perez-Encinas M, Ferrer-Marin F, Mata-Vazquez MI, Raya JM, Estrada N, Garcia S, Kerguelen A, Duran MA, Albors M, Cervantes F. Predictive factors for anemia response to erythropoiesis-stimulating agents in myelofibrosis. Eur J Haematol. 2017 Apr;98(4):407-414. doi: 10.1111/ejh.12846. Epub 2017 Jan 19. PMID 28009442
- [Background] Tefferi A, Cervantes F, Mesa R, Passamonti F, Verstovsek S, Vannucchi AM, Gotlib J, Dupriez B, Pardanani A, Harrison C, Hoffman R, Gisslinger H, Kroger N, Thiele J, Barbui T, Barosi G. Revised response criteria for myelofibrosis: International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus report. Blood. 2013 Aug 22;122(8):1395-8. doi: 10.1182/blood-2013-03-488098. Epub 2013 Jul 9. PMID 23838352
- [Background] Barosi G, Mesa R, Finazzi G, Harrison C, Kiladjian JJ, Lengfelder E, McMullin MF, Passamonti F, Vannucchi AM, Besses C, Gisslinger H, Samuelsson J, Verstovsek S, Hoffman R, Pardanani A, Cervantes F, Tefferi A, Barbui T. Revised response criteria for polycythemia vera and essential thrombocythemia: an ELN and IWG-MRT consensus project. Blood. 2013 Jun 6;121(23):4778-81. doi: 10.1182/blood-2013-01-478891. Epub 2013 Apr 16. PMID 23591792
- [Background] Tefferi A, Guglielmelli P, Larson DR, Finke C, Wassie EA, Pieri L, Gangat N, Fjerza R, Belachew AA, Lasho TL, Ketterling RP, Hanson CA, Rambaldi A, Finazzi G, Thiele J, Barbui T, Pardanani A, Vannucchi AM. Long-term survival and blast transformation in molecularly annotated essential thrombocythemia, polycythemia vera, and myelofibrosis. Blood. 2014 Oct 16;124(16):2507-13; quiz 2615. doi: 10.1182/blood-2014-05-579136. Epub 2014 Jul 18. PMID 25037629
- [Background] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger MW, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner EO, Lyons RM, Raza A, Vaddi K, Sun W, Peng W, Sandor V, Kantarjian H; COMFORT-I investigators. Efficacy, safety, and survival with ruxolitinib in patients with myelofibrosis: results of a median 3-year follow-up of COMFORT-I. Haematologica. 2015 Apr;100(4):479-88. doi: 10.3324/haematol.2014.115840. Epub 2015 Jan 23. PMID 25616577
- [Background] Newberry KJ, Patel K, Masarova L, Luthra R, Manshouri T, Jabbour E, Bose P, Daver N, Cortes J, Kantarjian H, Verstovsek S. Clonal evolution and outcomes in myelofibrosis after ruxolitinib discontinuation. Blood. 2017 Aug 31;130(9):1125-1131. doi: 10.1182/blood-2017-05-783225. Epub 2017 Jul 3. PMID 28674026
- [Background] Vannucchi AM, Guglielmelli P. Traffic lights for ruxolitinib. Blood. 2017 Aug 31;130(9):1075-1077. doi: 10.1182/blood-2017-07-795880. No abstract available. PMID 28860323
- [Background] Huang J, Tefferi A. Erythropoiesis stimulating agents have limited therapeutic activity in transfusion-dependent patients with primary myelofibrosis regardless of serum erythropoietin level. Eur J Haematol. 2009 Aug;83(2):154-5. doi: 10.1111/j.1600-0609.2009.01266.x. Epub 2009 Apr 10. No abstract available. PMID 19366369
- [Background] Akel S, Petrow-Sadowski C, Laughlin MJ, Ruscetti FW. Neutralization of autocrine transforming growth factor-beta in human cord blood CD34(+)CD38(-)Lin(-) cells promotes stem-cell-factor-mediated erythropoietin-independent early erythroid progenitor development and reduces terminal differentiation. Stem Cells. 2003;21(5):557-67. doi: 10.1634/stemcells.21-5-557. PMID 12968110
- [Background] Soderberg SS, Karlsson G, Karlsson S. Complex and context dependent regulation of hematopoiesis by TGF-beta superfamily signaling. Ann N Y Acad Sci. 2009 Sep;1176:55-69. doi: 10.1111/j.1749-6632.2009.04569.x. PMID 19796233
- [Background] Scandura JM, Boccuni P, Massague J, Nimer SD. Transforming growth factor beta-induced cell cycle arrest of human hematopoietic cells requires p57KIP2 up-regulation. Proc Natl Acad Sci U S A. 2004 Oct 19;101(42):15231-6. doi: 10.1073/pnas.0406771101. Epub 2004 Oct 11. PMID 15477587
- [Background] Brenet F, Kermani P, Spektor R, Rafii S, Scandura JM. TGFbeta restores hematopoietic homeostasis after myelosuppressive chemotherapy. J Exp Med. 2013 Mar 11;210(3):623-39. doi: 10.1084/jem.20121610. Epub 2013 Feb 25. PMID 23440043
- [Background] Chabanon A, Desterke C, Rodenburger E, Clay D, Guerton B, Boutin L, Bennaceur-Griscelli A, Pierre-Louis O, Uzan G, Abecassis L, Bourgeade MF, Lataillade JJ, Le Bousse-Kerdiles MC. A cross-talk between stromal cell-derived factor-1 and transforming growth factor-beta controls the quiescence/cycling switch of CD34(+) progenitors through FoxO3 and mammalian target of rapamycin. Stem Cells. 2008 Dec;26(12):3150-61. doi: 10.1634/stemcells.2008-0219. Epub 2008 Aug 28. PMID 18757300
- [Background] Zermati Y, Fichelson S, Valensi F, Freyssinier JM, Rouyer-Fessard P, Cramer E, Guichard J, Varet B, Hermine O. Transforming growth factor inhibits erythropoiesis by blocking proliferation and accelerating differentiation of erythroid progenitors. Exp Hematol. 2000 Aug;28(8):885-94. doi: 10.1016/s0301-472x(00)00488-4. PMID 10989189
- [Background] Zhou L, Nguyen AN, Sohal D, Ying Ma J, Pahanish P, Gundabolu K, Hayman J, Chubak A, Mo Y, Bhagat TD, Das B, Kapoun AM, Navas TA, Parmar S, Kambhampati S, Pellagatti A, Braunchweig I, Zhang Y, Wickrema A, Medicherla S, Boultwood J, Platanias LC, Higgins LS, List AF, Bitzer M, Verma A. Inhibition of the TGF-beta receptor I kinase promotes hematopoiesis in MDS. Blood. 2008 Oct 15;112(8):3434-43. doi: 10.1182/blood-2008-02-139824. Epub 2008 May 12. PMID 18474728
- [Background] Komrokji R, Garcia-Manero G, Ades L, Prebet T, Steensma DP, Jurcic JG, Sekeres MA, Berdeja J, Savona MR, Beyne-Rauzy O, Stamatoullas A, DeZern AE, Delaunay J, Borthakur G, Rifkin R, Boyd TE, Laadem A, Vo B, Zhang J, Puccio-Pick M, Attie KM, Fenaux P, List AF. Sotatercept with long-term extension for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes: a phase 2, dose-ranging trial. Lancet Haematol. 2018 Feb;5(2):e63-e72. doi: 10.1016/S2352-3026(18)30002-4. Epub 2018 Jan 10. PMID 29331635
- [Background] Platzbecker U, Germing U, Gotze KS, Kiewe P, Mayer K, Chromik J, Radsak M, Wolff T, Zhang X, Laadem A, Sherman ML, Attie KM, Giagounidis A. Luspatercept for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes (PACE-MDS): a multicentre, open-label phase 2 dose-finding study with long-term extension study. Lancet Oncol. 2017 Oct;18(10):1338-1347. doi: 10.1016/S1470-2045(17)30615-0. Epub 2017 Sep 1. PMID 28870615
- [Background] Zhang H, Kozono DE, O'Connor KW, Vidal-Cardenas S, Rousseau A, Hamilton A, Moreau L, Gaudiano EF, Greenberger J, Bagby G, Soulier J, Grompe M, Parmar K, D'Andrea AD. TGF-beta Inhibition Rescues Hematopoietic Stem Cell Defects and Bone Marrow Failure in Fanconi Anemia. Cell Stem Cell. 2016 May 5;18(5):668-81. doi: 10.1016/j.stem.2016.03.002. Epub 2016 Mar 24. PMID 27053300
- [Background] Herbertz S, Sawyer JS, Stauber AJ, Gueorguieva I, Driscoll KE, Estrem ST, Cleverly AL, Desaiah D, Guba SC, Benhadji KA, Slapak CA, Lahn MM. Clinical development of galunisertib (LY2157299 monohydrate), a small molecule inhibitor of transforming growth factor-beta signaling pathway. Drug Des Devel Ther. 2015 Aug 10;9:4479-99. doi: 10.2147/DDDT.S86621. eCollection 2015. PMID 26309397
- [Background] Badalucco S, Di Buduo CA, Campanelli R, Pallotta I, Catarsi P, Rosti V, Kaplan DL, Barosi G, Massa M, Balduini A. Involvement of TGFbeta1 in autocrine regulation of proplatelet formation in healthy subjects and patients with primary myelofibrosis. Haematologica. 2013 Apr;98(4):514-7. doi: 10.3324/haematol.2012.076752. Epub 2013 Feb 12. PMID 23403314
- [Background] Ciurea SO, Merchant D, Mahmud N, Ishii T, Zhao Y, Hu W, Bruno E, Barosi G, Xu M, Hoffman R. Pivotal contributions of megakaryocytes to the biology of idiopathic myelofibrosis. Blood. 2007 Aug 1;110(3):986-93. doi: 10.1182/blood-2006-12-064626. Epub 2007 May 1. PMID 17473062
- [Background] Gastinne T, Vigant F, Lavenu-Bombled C, Wagner-Ballon O, Tulliez M, Chagraoui H, Villeval JL, Lacout C, Perricaudet M, Vainchenker W, Benihoud K, Giraudier S. Adenoviral-mediated TGF-beta1 inhibition in a mouse model of myelofibrosis inhibit bone marrow fibrosis development. Exp Hematol. 2007 Jan;35(1):64-74. doi: 10.1016/j.exphem.2006.08.016. PMID 17198875
- [Background] Martyre MC, Romquin N, Le Bousse-Kerdiles MC, Chevillard S, Benyahia B, Dupriez B, Demory JL, Bauters F. Transforming growth factor-beta and megakaryocytes in the pathogenesis of idiopathic myelofibrosis. Br J Haematol. 1994 Sep;88(1):9-16. doi: 10.1111/j.1365-2141.1994.tb04970.x. PMID 7803262
- [Background] Zingariello M, Martelli F, Ciaffoni F, Masiello F, Ghinassi B, D'Amore E, Massa M, Barosi G, Sancillo L, Li X, Goldberg JD, Rana RA, Migliaccio AR. Characterization of the TGF-beta1 signaling abnormalities in the Gata1low mouse model of myelofibrosis. Blood. 2013 Apr 25;121(17):3345-63. doi: 10.1182/blood-2012-06-439661. Epub 2013 Mar 5. PMID 23462118
- [Background] Ponce CC, de Lourdes F Chauffaille M, Ihara SS, Silva MR. The relationship of the active and latent forms of TGF-beta1 with marrow fibrosis in essential thrombocythemia and primary myelofibrosis. Med Oncol. 2012 Dec;29(4):2337-44. doi: 10.1007/s12032-011-0144-1. Epub 2011 Dec 27. PMID 22200991
- [Background] Bock O, Loch G, Schade U, von Wasielewski R, Schlue J, Kreipe H. Aberrant expression of transforming growth factor beta-1 (TGF beta-1) per se does not discriminate fibrotic from non-fibrotic chronic myeloproliferative disorders. J Pathol. 2005 Apr;205(5):548-57. doi: 10.1002/path.1744. PMID 15726648
- [Background] Shehata M, Schwarzmeier JD, Hilgarth M, Hubmann R, Duechler M, Gisslinger H. TGF-beta1 induces bone marrow reticulin fibrosis in hairy cell leukemia. J Clin Invest. 2004 Mar;113(5):676-85. doi: 10.1172/JCI19540. PMID 14991065
- [Background] Ceglia I, Dueck AC, Masiello F, Martelli F, He W, Federici G, Petricoin EF 3rd, Zeuner A, Iancu-Rubin C, Weinberg R, Hoffman R, Mascarenhas J, Migliaccio AR. Preclinical rationale for TGF-beta inhibition as a therapeutic target for the treatment of myelofibrosis. Exp Hematol. 2016 Dec;44(12):1138-1155.e4. doi: 10.1016/j.exphem.2016.08.007. Epub 2016 Aug 31. PMID 27592389
- [Background] Margolskee E, Krichevsky S, Orazi A, Silver RT. Evaluation of bone marrow morphology is essential for assessing disease status in recombinant interferon alpha-treated polycythemia vera patients. Haematologica. 2017 Mar;102(3):e97-e99. doi: 10.3324/haematol.2016.153973. Epub 2016 Nov 3. No abstract available. PMID 27810993
- [Background] Anand S, Stedham F, Beer P, Gudgin E, Ortmann CA, Bench A, Erber W, Green AR, Huntly BJ. Effects of the JAK2 mutation on the hematopoietic stem and progenitor compartment in human myeloproliferative neoplasms. Blood. 2011 Jul 7;118(1):177-81. doi: 10.1182/blood-2010-12-327593. Epub 2011 May 11. PMID 21562050
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Scherber R, Dueck AC, Johansson P, Barbui T, Barosi G, Vannucchi AM, Passamonti F, Andreasson B, Ferarri ML, Rambaldi A, Samuelsson J, Birgegard G, Tefferi A, Harrison CN, Radia D, Mesa RA. The Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF): international prospective validation and reliability trial in 402 patients. Blood. 2011 Jul 14;118(2):401-8. doi: 10.1182/blood-2011-01-328955. Epub 2011 May 2. PMID 21536863
- [Background] Mascarenhas J, Hoffman R, Talpaz M, Gerds AT, Stein B, Gupta V, Szoke A, Drummond M, Pristupa A, Granston T, Daly R, Al-Fayoumi S, Callahan JA, Singer JW, Gotlib J, Jamieson C, Harrison C, Mesa R, Verstovsek S. Pacritinib vs Best Available Therapy, Including Ruxolitinib, in Patients With Myelofibrosis: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):652-659. doi: 10.1001/jamaoncol.2017.5818. PMID 29522138
- [Background] Harrison C, Kiladjian JJ, Al-Ali HK, Gisslinger H, Waltzman R, Stalbovskaya V, McQuitty M, Hunter DS, Levy R, Knoops L, Cervantes F, Vannucchi AM, Barbui T, Barosi G. JAK inhibition with ruxolitinib versus best available therapy for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):787-98. doi: 10.1056/NEJMoa1110556. PMID 22375970

RESULTS

PARTICIPANT FLOW:
Groups:
- Vacosertib 50 mg BID: Vactosertib intra-patient dose finding cohort.
  Vactosertib: 50 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
- Vacosertib 100 mg BID: Vactosertib: 100 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
- Vacosertib 150 mg BID: Vactosertib: 150 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
- Vacosertib 200mg BID: Vactosertib: 200 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
- Tier 2: Vactosertib: This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
Period: Vactosertib 50 mg BID (Tier 1)
Arm/Group | Vacosertib 50 mg BID | Vacosertib 100 mg BID | Vacosertib 150 mg BID | Vacosertib 200mg BID | Tier 2: Vactosertib
Started | 2 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Vactosertib 100 mg BID (Tier 1)
Arm/Group | Vacosertib 50 mg BID | Vacosertib 100 mg BID | Vacosertib 150 mg BID | Vacosertib 200mg BID | Tier 2: Vactosertib
Started | 0 | 2 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Vactosertib 150 mg BID (Tier 1)
Arm/Group | Vacosertib 50 mg BID | Vacosertib 100 mg BID | Vacosertib 150 mg BID | Vacosertib 200mg BID | Tier 2: Vactosertib
Started | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Vactosertib 200 mg BID (Tier 1)
Arm/Group | Vacosertib 50 mg BID | Vacosertib 100 mg BID | Vacosertib 150 mg BID | Vacosertib 200mg BID | Tier 2: Vactosertib
Started | 0 | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Vactosertib (Tier 2)
Arm/Group | Vacosertib 50 mg BID | Vacosertib 100 mg BID | Vacosertib 150 mg BID | Vacosertib 200mg BID | Tier 2: Vactosertib
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Vactosertib intra-patient dose finding cohort.
  Vactosertib This drug is a TG-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Identify the Safest, Minimally Effective Starting Dose Level for Patients on Tier 1
Description: The safest minimally effective dose is defined as the lowest dose level for which no dose limiting toxicity (DLT) was observed in Tier 1 AND the lowest dose level for which at least one of the 12 subjects enrolled on Tier 1 meet Criteria for Clinical Benefit
Time Frame: Baseline to week 16
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 2
mg | 50

2. Primary Outcome: Identify Dose Limiting Toxicities (DLTs) in Patients With MPN Enrolled on Tier 1
Description: Identify the incidence of dose limiting toxicity (DLT) within the first 12 weeks which are defined as:
  1. Any non-hematologic grade ≥3 toxicity except for nausea, vomiting or diarrhea lasting 3 days or less
  2. Any grade 4 neutropenia of any duration
  3. Any grade ≥3 neutropenia that has not recovered to grade ≥2 within 7 days of onset
  4. Any grade ≥3 febrile neutropenia
  5. Any grade ≥3 thrombocytopenia associated with clinically significant bleeding or requiring platelet transfusion
Time Frame: Baseline to week 12
Measure: Number; unit: Count of DLTs
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200mg BID
Number analyzed (Participants) | 2 | 2 | 2 | 2
Count of DLTs | 0 | 0 | 0 | 0

3. Primary Outcome: Identify the Maximum Tolerated Dose (MTD) of Vactosertib in Patients With MPN Enrolled on Tier 1
Description: Identify the Maximum Tolerated Dose (MTD) of vactosertib defined as the highest dose which does not meet the Tier 1 stopping rule. The tier 1 stopping rule is triggered if any patient experiences a Grade 5 dose limiting toxicity within the first 12 weeks of starting vactosertib or if more than five patients experience a dose limiting toxicity at any dose within the first 12 weeks on study.
Time Frame: Baseline to week 12
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 2
mg | 200

4. Primary Outcome: Number of Tier 2 Patients Who Have Achieved Erythropoietic Response as Defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Criteria
Description: Number of patients who achieve an erythropoietic response defined by:
  1. HGB increase of 1.5g/dL compared to baseline hemoglobin;
  2. Reduction in PRBC transfusion rate to ≤ 50% of pre-treatment transfusion rate; or
  3. Reduction in PRBC transfusions by ≥ 4 Units over an 8-week period.
Time Frame: baseline to week 16
Population: No subjects went on to the Tier 2 portion of the study
Groups:
- Tier 2: Vactosertib: Vactosertib This drug is a TG-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
Arm/Group | Tier 2: Vactosertib
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Tier 2 Patients Who Have Achieved Clinical Response in Symptoms as Defined by International Working Group (IWG) Criteria
Description: Number of patients who have achieved clinical response defined by a reduction in Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) total score by ≥ 50% compared to pretreatment score
Time Frame: baseline to week 16
Population: No subjects went on to the Tier 2 portion of the study
Arm/Group | Tier 2: Vactosertib
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Tier 2 Patients Who Have Achieved Splenic Response in Symptoms as Defined by International Working Group (IWG) Criteria
Description: Number of patients who have achieved splenic response defined by:
  1. Non-palpable spleen when baseline spleen size was 5-10 cm below left costal margin;
  2. At least 50% reduction in spleen size when baseline spleen is > 10 cm below left costal margin
  3. At least 35% reduction in spleen size as assessed by US, CT or MRI.
Time Frame: baseline to week 16
Population: No subjects went on to the Tier 2 portion of the study
Arm/Group | Tier 2: Vactosertib
Number analyzed (Participants) | 0

7. Primary Outcome: Identify Dose Limiting Toxicities (DLTs) in Patients With MPN Enrolled on Tier 2
Description: Identify the number of dose limiting toxicities (DLT) within the first 12 weeks which are defined as:
  1. Any non-hematologic grade ≥3 toxicity except for nausea, vomiting or diarrhea lasting 3 days or less
  2. Any grade 4 neutropenia of any duration
  3. Any grade ≥3 neutropenia that has not recovered to grade ≥2 within 7 days of onset
  4. Any grade ≥3 febrile neutropenia
  5. Any grade ≥3 thrombocytopenia associated with clinically significant bleeding or requiring platelet transfusion
Time Frame: baseline to week 12
Population: No subjects went on to the Tier 2 portion of the study
Arm/Group | Tier 2: Vactosertib
Number analyzed (Participants) | 0

8. Primary Outcome: Identify the Maximum Tolerated Dose (MTD) of Vactosertib in Patients With MPN Enrolled on Tier 2
Description: Identify the Maximum Tolerated Dose (MTD) of vactosertib defined as the highest dose which does not meet the Tier 2 stopping rule. The tier 2 stopping rule is triggered if any patient experiences a Grade 5 dose limiting toxicity within the first 12 weeks of starting vactosertib or if more than five patients experience a dose limiting toxicity at any dose within the first 12 weeks on study.
Time Frame: baseline to week 12
Population: No subjects went on to the Tier 2 portion of the study
Arm/Group | Tier 2: Vactosertib
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Patients in Which a Histological Response is Seen
Description: Histological response is defined by reduction of any amount in grade of bone marrow fibrosis by histopathologic assessment at 16 weeks.
Time Frame: 16 weeks
Population: 0 subjects were analyzed for Tier 1 subjects taking 50mg, 100mg, and 150mg of Vactosertib because no participants were taking those doses at 16 weeks. 0 subjects were analyzed in Tier 2 because no subjects were in Tier 2 at 16 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Tier 1: Vactosertib 50 mg BID: Vactosertib intra-patient dose finding cohort.
  Vactosertib: 50 mg BID This drug is a TG-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
- Tier 2: Vactosertib: This drug is a TG-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200mg BID | Tier 2: Vactosertib
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 0
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Patients in Which a Molecular Response is Seen
Description: Number of patients in which a molecular response is seen. Molecular response is defined by a decrease in VAF of MPN-driver mutations (eg. JAK2, CALR, and MPL allelic ratio) in blood and/or bone marrow cells
Time Frame: 16 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200mg BID | Tier 2: Vactosertib
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 0
Participants | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Patients in Which a Pharmacodynamic Response is Seen
Description: A pharmacodynamic response is defined as any of the following:
  1. Reduced immunohistochemical staining for SMAD2/3 phosphorylation in bone marrow biopsy sections.
  2. Reduced mean fluorescence intensity of SMAD2/3 phosphorylation staining in peripheral blood hematopoietic stem and progenitor cells (HSPCs) or mature progeny as assessed by flow cytometry.
  3. Reduced mean fluorescence intensity of SMAD2/3 phosphorylation staining in bone marrow hematopoietic stem and progenitor cells (HSPCs) or mature progeny as assessed by flow cytometry.
Time Frame: 16 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200mg BID | Tier 2: Vactosertib
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 0
Participants | 0 | 0 | 0 | 1 | 0

12. Secondary Outcome: Number of Patients Who Have Experienced Any of the Following: Hematologic Toxicities, Infections, Disease Progression, and Thrombosis Events
Time Frame: baseline to 16 weeks
Population: No subjects enrolled on Tier 2
Measure: Count of Participants; unit: Participants
Groups:
- Tier 1: Vactosertib 200 mg BID: Vactosertib: 200 mg BID This drug is a TGF-Beta receptor type 1 inhibitor, by inhibiting phosphorylation of the ALK5 substrates SMAD2 and SMAD3. This inhibition could promote regeneration of normal human stem cells and proliferation of erythroid progenitors to treat the underlying hypoproliferative anemia in advanced MPNs.
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200 mg BID | Tier 2: Vactosertib
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 0
Participants | 0 | 0 | 1 | 2 | 0

13. Secondary Outcome: Overall Survival Defined as the Amount of Time a Patient is Alive After Starting Study Treatment
Description: The overall survival range describes the average length of time subjects were followed for survival
Time Frame: Week 1 Day 1 to 6 months post treatment discontinuation. This collection period for both subjects on study was over an average duration of 54 weeks.
Measure: Mean (Full Range); unit: Weeks
Arm/Group | All Participants
Number analyzed (Participants) | 2
Weeks | 54 [54 to 54]

14. Secondary Outcome: Progression Free Survival Defined as the Duration of Time From Start of Treatment to Time of Progression
Time Frame: Week 1 Day 1 to 6 months post treatment discontinuation
Measure: Mean (Full Range); unit: Weeks
Arm/Group | All Participants
Number analyzed (Participants) | 2
Weeks | 25.5 [21 to 30]

ADVERSE EVENTS:
Time Frame: Deaths were collected from Week 1 Day 1 through 6 months post treatment discontinuation. This collection period for both subjects on study was over an average duration of 54 weeks. Serious and Other (Not Including Serious) Adverse Events were collected while subjects were on treatment. This collection period for both subjects on study was over an average duration of 28 weeks.
Description: All subjects treated with Vactosertib
Arm/Group | Tier 1: Vactosertib 50 mg BID | Tier 1: Vactosertib 100 mg BID | Tier 1: Vactosertib 150 mg BID | Tier 1: Vactosertib 200mg BID | Tier 2: Vactosertib | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 0/0 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tier 1: Vactosertib 50 mg BID (N=2) | Tier 1: Vactosertib 100 mg BID (N=2) | Tier 1: Vactosertib 150 mg BID (N=2) | Tier 1: Vactosertib 200mg BID (N=2) | Tier 2: Vactosertib (N=0) | All Participants (N=2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain extremity (left lower leg) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Only a small number of subjects was analyzed due to low accrual and early termination. Additionally, only Tier 1 outcome measures could be analyzed due to 0 subjects enrolling onto Tier 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT04103645/Prot_SAP_000.pdf